CLINICAL TRIAL: NCT03429907
Title: An Early Stress-Reduction Intervention in Patients With Newly Diagnosed Breast Cancer: A Randomized Pilot Study
Brief Title: An Early Stress-Reduction Intervention in Patients With Newly Diagnosed Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Hackett Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-0600; NCI-2018-01079 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2018-01-24; First posted 2018-02-12 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Malignant Neoplasm of Breast
Keywords: Malignant neoplasm of breast; Mind-Body Exercises; Questionnaires; Surveys
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mind-Body Exercises (Experimental): Participants do daily mind-body exercises for 14 days before starting chemotherapy. The exercises are presented on an online application ("app") that runs on participant's personal electronic device (such as a mobile phone or tablet).
  Questionnaires completed at baseline, at third and at last cycle of chemotherapy, and 6 months after chemotherapy.
  Interventions: Behavioral: Mind-Body Exercises; Behavioral: Questionnaires
- Standard of Care (Other): Questionnaires completed at baseline, at third and at last cycle of chemotherapy, and 6 months after chemotherapy.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Mind-Body Exercises — Participants do daily mind-body exercises for 14 days before starting chemotherapy. The exercises are about 10 minutes per day.
  Arms: Mind-Body Exercises
Behavioral: Questionnaires — Questionnaires completed at baseline, at third and at last cycle of chemotherapy, and 6 months after chemotherapy.
  Other Names: Surveys

SUMMARY:
The goal of this research study is to learn if starting a stress-reduction program before treatment can affect your stress, mood, and physical symptoms during and after treatment for cancer.

This is an investigational study.

Up to 140 participants will be enrolled in this study. All participants will be recruited at MD Anderson.

DETAILED DESCRIPTION:
Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. You will have an equal chance of being in either group:

* If you are in Group 1, you will be asked to do daily mind-body exercises for 14 days, beginning before you start receiving chemotherapy. The exercises are short, about 10 minutes per day. The exercises are presented on an online application ("app") that runs on your personal electronic device (such as a mobile phone or tablet). You will be required to install the application on your personal device and to create an account. The study staff will tell you how to perform the exercises, install the application, and create an account. During the 14 days, you will receive automated daily reminders to do the exercises. After you have finished the 14 days of mind-body exercises, you may continue to use the application free of charge for the remainder of the year. After the first year, if you want to keep using the application, you will have to pay for it.
* If you are in Group 2, you will not perform the mind-body exercises. You will be offered one year of free access to the application described above at your last study visit.

Study Visits - All Participants:

Before you start chemotherapy:

* You will complete 10 questionnaires about your stress, mood, physical symptoms, and personality. It should take about 45 minutes to complete all of the questionnaires. You can decide to complete some of the questionnaires from home on a personal computer.
* Information about you (such as age and race) and the disease will be collected from your medical record.
* Blood (about 1 tablespoon) will be drawn for testing of genes and biomarkers that may be related to physical symptoms and mood. Biomarkers are found in the blood and tissue and may help researchers measure the effects of the daily mind-body exercises.
* A hair sample will be taken to measure hormones that are commonly released during times of stress. A lock of hair about the width of a pencil lead will be cut close to your scalp.
* You may be asked to complete a computer task in which you press buttons multiple times in a set time limit. You will receive written instructions on how to complete the task. It should take 15 minutes to complete this task.

At about 15 days after you started the study:

°You will complete one question about your stress. You can complete this question in the clinic or from home on a personal computer.

During chemotherapy:

At about the third month and the sixth month of chemotherapy:

* You will complete 6 questionnaires about your stress, mood, and physical symptoms. It should take about 30 minutes to complete the questionnaires. You can decide to complete these questionnaires from home on a personal computer.
* If your schedule allows for it and you agree, blood (about 1 tablespoon) will be drawn for biomarker testing. If you do not have time to complete this blood draw, it will not affect your participation in this study.

About 6 months after you finish receiving chemotherapy:

* You will complete 8 questionnaires about your stress, mood, and physical symptoms. It should take about 30 minutes to complete the questionnaires.
* Blood (about 1 tablespoon) will be drawn for biomarker testing.
* You may be asked to complete the computer task described above.

Length of Study:

Your participation on this study will be over about 6 months after your last cycle of chemotherapy. If chemotherapy will not be the first treatment you receive for your diagnosis, then your participation on this study will be over at 2 weeks after the start of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Women with stage I-III breast cancer who are followed by the Department of Breast Medical Oncology and are recommended for neoadjuvant chemotherapy, any regimen. If chemotherapy is received in an outside facility, patients are eligible if they are scheduled to return to MD Anderson after completion of chemotherapy.
2. Patients = or > 18 years old
3. Patients who speak English
4. Patients who are willing and able to review, understand, and provide written consent
5. Patients who agree to comply with all study procedures
6. Patients who have access to a mobile phone, tablet, or personal computer, that supports the Headspace application

Exclusion Criteria:

1. Patients with a documented diagnosis of a formal thought disorder (e.g., schizophrenia)
2. Patients who are currently or have been in the past three months actively engaged in meditation-related exercises for at least one hour a week
3. Patients who are currently receiving psychotherapy
4. Patients with pre-existing diagnosis of an inflammatory autoimmune disease such as rheumatoid arthritis, systemic lupus erythematosus, or multiple sclerosis
5. Patients who are currently taking adrenergic receptor antagonist (e.g., propranolol) or corticosteroids (e.g., dexamethasone, methylprednisolone)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Effect of the Stress-Reduction Intervention on Changes in Patient-Reported Outcomes From T0 to T2 and T3 | Baseline up to 6 months after chemotherapy
  For the primary objective, changes from T0 to T2 and T3 in neurotoxic somatic symptoms analyzed with multilevel models, in which changes over time are estimated simultaneously across groups.

SECONDARY OUTCOMES:
Changes in Inflammatory Markers | Baseline up to 6 months after chemotherapy
  To determine the associations of patient-reported outcomes with inflammatory biomarkers, researchers will analyze parallel growth patterns in which correlations between intercept/slope in the PROs and intercept/slope in the biomarkers are tested.
  Cortisol assessed in hair samples. In vitro determination of the sensitivity of leukocytes for regulation by cortisol . Blood drawn for plasma levels of biomarkers of immunological activity (C-reactive protein (CRP), IL-6, soluble IL-6 receptor (sIL-6R) TNF-alpha, TNF-receptors I and II (TNF-RI and TNF-RII), and IL-1 receptor antagonist (IL-1RA)), and DAMPs (HSP70, HMGB1, sRAGE). Blood for assessment of cytokine levels in supernatants. Supernatants from T-cells stimulated with anti CD3 and anti CD28 assessed for levels of gamma-interferon, IL-2, IL-10, and IL4. Supernatants from monocytes stimulated with lipopolysaccharide assessed for levels of TNF-alpha and IL-10.
Associations of patient-reported stress and neuroendocrine biomarkers | Baseline up to 6 months after chemotherapy
  Described using cross-sectional Pearson's r correlations and multiple regression models including identified confounding variables.
  Cortisol assessed in hair samples. This measure will give insight into the amount of stress experienced in the past month, the time during which the participant was dealing with diagnostic tests and a possible breast cancer diagnosis.
Associations of patient-reported neurotoxic somatic and depressive symptoms with inflammatory biomarkers and mitochondrial functioning during and after chemotherapy. | Baseline up to 6 months after chemotherapy
  Blood for plasma levels of biomarkers of immunological activity (C-reactive protein (CRP), IL-6, soluble IL-6 receptor (sIL-6R) TNF-alpha, TNF-receptors I and II (TNF-RI and TNF-RII), and IL-1 receptor antagonist (IL-1RA)), and DAMPs (HSP70, HMGB1, sRAGE). Blood collected for analysis of mitochondrial function.
Determine the relation between motivational effort expenditure and the neurotoxic symptom fatigue. | Baseline up to 6 months after chemotherapy
  The ratio of high effort/low effort choices on the EEfRT analyzed with Generalized Estimating Equations (GEE) models, which allow for controlling for time-varying covariates such as trial number.
The association between EEfRT outcome and patient-reported stress and personality characteristics assessed with separate GEE models | Baseline up to 6 months after chemotherapy
Changes in Mitochondrial Function | Baseline up to 6 months after chemotherapy
  To determine the associations of patient-reported outcomes with mitochondrial function, researchers will analyze parallel growth patterns in which correlations between intercept/slope in the PROs and intercept/slope in the biomarkers are tested.

CONTACTS AND LOCATIONS:
Overall Officials: Keri Schadler, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org